CLINICAL TRIAL: NCT05042973
Title: Empagliflozin to Elderly and Obese Patients With Cardiovascular Disease (Empire Prevent: Metabolic): A Randomized Controlled Trial
Brief Title: The Metabolic Effects of Empagliflozin in Patients With High Risk of Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jacob Moller (Other)
Collaborators: Danish Heart Foundation (Other); Herlev and Gentofte Hospital (Other); University Hospital Bispebjerg and Frederiksberg (Other); Hillerod Hospital, Denmark (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor-Investigator, Jacob Moller, Professor, MD, PhD, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: S-20210028-2
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Obesity; Heart Failure
Keywords: Renal function; Glucose intolerance; Lipid metabolism
MeSH Terms: conditions — Obesity; Heart Failure; Glucose Intolerance | interventions — empagliflozin

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active drug (Empagliflozin) (Active Comparator): Empagliflozin 10 mg, 1 capsule per day
  Interventions: Drug: Empagliflozin 10 MG
- Inactive drug (placebo) (Placebo Comparator): Placebo, 1 capsule per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin 10 MG — Patients are randomized 1:1 to receive either Empagliflozin or matching placebo for 180 days
  Arms: Active drug (Empagliflozin)
Drug: Placebo — Placebo matches the active drug in appearance, odor and labelling.
  Arms: Inactive drug (placebo)

SUMMARY:
The aim of this trial is to assess the effect of Empagliflozin on lipid and glucose metabolism as well as volume homeostasis and renal function in elderly and obese patients with increased risk of developing heart failure. No history of established heart failure or diabetes is allowed.

The primary hypotheses are that 6 months treatment with Empagliflozin 10 mg a day will: 1) decrease epicardial adipose tissue volume, and 2) reduce estimated extracellular volume compared with placebo.

DETAILED DESCRIPTION:
The Empire Prevent: Metabolic is a part of the Empire Prevent Trial Program, which also comprises the Empire Prevent: Cardiac.

The Empire Prevent: Metabolic is designed to enroll at least 120 patients.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index >28kg/m2
* Age 60-84 years
* Established risk factor for developing heart failure, defined as at least one of the following:
* hypertension
* ischemic heart disease
* stroke/transient cerebral ischemia
* chronic kidney disease (eGFR 30-45ml/min/1.73m2)

Exclusion Criteria:

* Diabetes mellitus type 1 or 2 (no medical history, no antidiabetic treatment)
* Heart failure with reduced ejection fraction (LVEF <40%)
* Inability to perform exercise test
* Dementia
* Severe non-compliance
* Substance abuse
* Severe chronic obstructive pulmonary disease (FEV1<50% expected value)
* Permanent atrial fibrillation
* GFR <30 ml/min/1,73m2
* Severe peripheral artery disease
* Cancer treatment within one year beside prostate cancer and basal cell carcinoma
* Severe aortic or mitral valve disease
* Pregnancy or breastfeeding
* Acute hospital admission within 30 days
* Participation in other pharmacological study

Ages: 60 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2025-01-16 (Actual); Study Completion 2025-01-23 (Actual)

PRIMARY OUTCOMES:
Ventricular epicardial adipose tissue (EAT) mass | 180 days
  Between-group difference in the change of EAT mass assessed by cardiac magnetic resonance imaging (MRI)
Estimated extracellular volume (eECV) | 180 days
  Between-group difference in the change of eECV assessed by 99mTc-DTPA clearance (technetium-99mTc-diethylenetriaminepentaacetic acid)

SECONDARY OUTCOMES:
Total pericardial adipose tissue volume | 180 days
  Between-group difference in the change of pericardial adipose tissue volume assessed by cardiac MRI
Total epicardial adipose tissue (EAT) volume | 180 days
  Between-group difference in the change of EAT mass assessed by cardiac magnetic resonance imaging (MRI)
Plasma volume | 180 days
  Between-group difference in the change of estimated plasma volume assessed by hematocrit and hemoglobin
Right ventricular end-diastolic volume index, RVEDVI | 180 days
  Between-group difference in the change of RVEDVI assessed by cardiac MRI

OTHER OUTCOMES:
Erythropoietin | 180 days
  Between-group difference in the change of erythropoietin
Exploratory outcome: fat tissue gene expression | 180 days
  Between-group difference in fat tissue gene expression assessed by Western Blot
Exploratory outcome: oxidative stress and inflammation. | 180 days
  Between-group difference in biomarkers of oxidative stress and inflammation.
Ketone bodies | 180 days
  Between-group difference in the change of ketone supply to the heart assessed by blood ketones
Urine albumin/creatinine ratio | 180 days
  Between-group difference in the change of urine albumin/creatinine ratio
Uric acid | 180 days
  Between-group difference in the change of uric acid
Kidney function (estimated) | 180 days
  Between-group difference in the change of estimated glomerular filtration rate (eGFR) based on the chronic kidney disease epidemiology collaboration (CKD-EPI) estimation
Kidney function (measured) | 180 days
  Between-group difference in the change of glomerular filtration rate assessed by 99mTc-DTPA clearance
Glucose tolerance | 180 days
  Between-group difference in the change of glucose metabolism assessed by oral glucose tolerance test
Body composition | 180 days
  Between-group difference in the change in body composition assessed by dual energy x-ray absorptiometry (DXA) scan

CONTACTS AND LOCATIONS:
Overall Officials: Morten Schou, MD, PhD, Principal Investigator — Herlev-Gentofte Hospital; Jacob Eifer Møller, MD, PhD, Principal Investigator — Odense University Hospital
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Andersen CF, Larsen JH, Jensen J, Omar M, Nouhravesh N, Kistorp C, Tuxen C, Gustafsson F, Knop FK, Forman JL, Davidovski FS, Jensen LT, Hojlund K, Kober L, Antonsen L, Poulsen MK, Schou M, Moller JE. Empagliflozin to elderly and obese patients with increased risk of developing heart failure: Study protocol for the Empire Prevent trial program. Am Heart J. 2024 May;271:84-96. doi: 10.1016/j.ahj.2024.02.005. Epub 2024 Feb 15. PMID 38365073

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-01-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT05042973/SAP_000.pdf